# **Effect of Beetroot Extract Supplementation on the Athletic Performance of Trained Rugby Athletes**

### NCT07106489

Last version: January 15, 2025

## Effect of Beetroot Extract Supplementation on the Athletic Performance of Trained Rugby Athletes.

This document is divided into two parts: first, the information related to the project, and then the consent form for each participant. Thus, by signing this document, each participant agrees to participate in the study, and the researchers agree to comply with the terms described in here

#### Justification:

In the field of sports, sports supplementation has gained great importance for improving athletic performance, which is why research on this topic continues. In recent years, nitrate supplementation (from foods rich in these compounds, such as beetroot) has been widely studied, finding benefits in various sports. However, their studies have focused on cyclical sports (such as endurance, cycling, swimming, etc.), and little research has been found on no cyclical sports (such as ball sports, including rugby), and current studies are inconclusive regarding their effect on these sports, highlighting the importance of conducting research in this area.

#### **Objective:**

To establish the effect of nitrate-rich beetroot extract supplementation on the athletic performance of rugby players. To achieve this objective, we seek to determine whether supplementation has an effect on various physical skills necessary in team sports, such as acceleration, speed, and strength.

#### Description of the study, procedure, and purpose:

Participants in the study who provide their consent and meet the required criteria will participate. Initially, a nutritional assessment will be conducted, which includes the collection of personal and socioeconomic data and questionnaires to identify food consumption, as well as an anthropometric assessment (the results of which will be provided to each athlete). The physical tests to be performed are listed below:

- 1. 40-meter test
- 2. Bronco test
- 3. Back squat
- 4. Chest press

A questionnaire will also be administered to identify the perception of fatigue, known as the Borg scale.

#### Discomfort or risks during participation:

The research is classified as minimal risk because no high-risk procedures will be performed. However, professionals in each area are available to ensure the necessary precautions are taken and minimize any discomfort that may occur.

#### Benefits that may be obtained:

During the study, a complete nutritional evaluation with corresponding counseling will be obtained, which can be useful for the athlete to improve both, their health and athletic performance. In addition, the anthropometric results are also useful in other areas related to health and performance.

#### **Questions and information:**

Any updated information discovered during the study will be duly informed, even if it may affect your willingness to continue participating. Additionally, if you have any questions or require clarification regarding procedures, risks, benefits, and anything else related to the research, you can contact researcher Leidy Tatiana Reyes Vega at 301 697 1711 or at Itreyesv@unal.edu.co. Responses are not limited to electronic means; if you wish to ask the researcher questions in person during the research, you are committed to providing the requested information.

#### Participation/Voluntary Withdrawal:

Your participation is entirely voluntary, so you are free to withdraw your consent at any time and cease participating without prejudice or penalty. Furthermore, the researcher may also withdraw participation if deemed appropriate, and the reasons for this will be fully documented.

#### **Confidentiality and Privacy:**

The information, measurements, and data collected during the study will be treated confidentially. The publication of the results guarantees privacy, so each participant will not be identified. The results to be delivered will be shared only personally with each participant. Likewise, the use of the acquired data for future projects and/or research is authorized, without affecting the confidentiality and privacy of the participants.

| l, | , identified with ID: CC CE P1 |
|---|---|
| ,number | , have read and understand this document and have no |
| • • | ntent, since I have had the opportunity to ask questions and be<br>untarily consent to authorize the research. |
| Signature: | Email: |
| Date: | Phone: |